CLINICAL TRIAL: NCT04988217
Title: A Phase I/II Randomized, Double-blind, Placebo-controlled Study of Inhaled Interferon α2b for the Treatment of Coronavirus Disease 19 (COVID-19)
Brief Title: Inhaled Interferon α2b for the Treatment of Coronavirus Disease 19 (COVID-19)
Acronym: IN2COVID
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Pontificia Universidad Catolica de Chile (Other)
Collaborators: Altum Pharmaceuticals INC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 210224003
Record Dates: First submitted 2021-07-22; First posted 2021-08-03 (Actual); Last update posted 2022-08-05 (Actual); Status verified 2022-04

CONDITIONS: Coronavirus Disease 2019
Keywords: Interferon alpha 2b; COVID-19
MeSH Terms: conditions — COVID-19 | interventions — Interferon-alpha2b

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Part 1a: Interferon alpha 2b 2.5 MIU (Experimental): Nebulized interferon alpha 2b 2.5 MIU every 12 hours during 10 days (20 doses total)
  Interventions: Drug: Interferon-Alpha2B
- Part 1b: Interferon alpha 2b 5 MIU (Experimental): Nebulized interferon alpha 2b 5 MIU every 12 hours during 10 days (20 doses total)
  Interventions: Drug: Interferon-Alpha2B
- Part 1: Placebo (Placebo Comparator): Nebulized placebo every 12 hours during 10 days (20 doses total)
  Interventions: Drug: Placebo
- Part 2: Interferon alpha 2b 5 MIU (or maximum tolerated dose from part 1) (Experimental): Nebulized interferon alpha 2b 5 MIU (or maximum tolerated dose from part 1) every 12 hours during 10 days (20 doses total)
  Interventions: Drug: Interferon-Alpha2B
- Part 2: Placebo (Placebo Comparator): Nebulized placebo every 12 hours during 10 days (20 doses total)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Interferon-Alpha2B — Nebulized interferon alpha 2B
  Other Names: AP-003
  Arms: Part 1a: Interferon alpha 2b 2.5 MIU; Part 1b: Interferon alpha 2b 5 MIU; Part 2: Interferon alpha 2b 5 MIU (or maximum tolerated dose from part 1)
Drug: Placebo — Nebulized placebo
  Arms: Part 1: Placebo; Part 2: Placebo

SUMMARY:
The IN2COVID Study is a 2-staged phase I/II double-blind, randomized, placebo-controlled trial to evaluate the efficacy and safety of AP-003 (Interferon α2b) when administered via inhalation twice daily for 10 days. Participants will have a final visit at Day 11.

A lead-in phase 1 substudy will be performed with at least 18 healthy adult male subjects to assess safety and tolerability of inhaled AP-003 compared to placebo for 10 days. Two cohorts of 9 subjects will be randomly assigned to receive two doses of inhaled AP-003 or placebo with an allocation ratio of 2:1. The first cohort will assess a dose of 2.5 MIU of inhaled AP-003. If no adverse events are observed, the second cohort will be conducted using a dose of 5 MIU of inhaled AP-003. Maximum tolerated dose will be determined in this phase 1 substudy.

After the completion of phase 1, the study will continue with a phase 2 treatment RCT in patients with COVID-19. In this phase, 150 adults with mild or moderate COVID-19 demonstrated by SARS-CoV-2 positive polymerase chain reaction (PCR) ≤ 5 days at enrollment will be randomized 1:1 (75 in each arm) to receive nebulized AP-003 or identical placebo twice daily during 10 days.

ELIGIBILITY:
Phase 1 stage:

Inclusion criteria:

1. Male subjects aged 18-50 years;
2. In good state of health, determined by medical history, physical exam, and normal laboratory tests at screening;
3. Are able to provide informed consent for participation;
4. Are able and willing to comply with the study schedule and procedures.

Exclusion Criteria

1. Active SARS-CoV-2 infection demonstrated by positive polymerase chain reaction (PCR) at enrollment;
2. Requiring CPAP for sleep apnea;
3. Pre-existing pulmonary disease;
4. Have any serious acute concomitant illness that, in the opinion of the investigator, would interfere with evaluation of safety of AP-003, or put the participant at risk of harm from study participation;
5. Are currently receiving an investigational agent, have participated in another study of an investigational agent within 30 days of enrollment, or were previously enrolled in the current study;
6. Are legally incompetent and unable to understand the study's purpose, significance, and consequences, and to make decisions accordingly;
7. Have known hypersensitivity to interferon alpha or any component of the study drug or placebo control.

Phase 2 stage:

Inclusion criteria:

1. Active SARS-CoV-2 infection demonstrated by positive polymerase chain reaction (PCR) ≤ 5 days at enrollment;
2. Symptomatic of mild or moderate COVID-19 for ≤ 5 days at enrollment. Symptoms can include fever, cough, sore throat, malaise, headache, muscle pain, gastrointestinal symptoms, chest pain, with or without shortness of breath on exertion/dyspnea;
3. Age ≥ 18 years;
4. Are able to provide informed consent for participation;
5. Are able and willing to comply with the study schedule and procedures.

Exclusion Criteria

1. Patients requiring CPAP for sleep apnea.
2. Patients with pre-existing pulmonary disease requiring chronic O2 supplementation.
3. Patients with known infection with Influenza A or B;
4. In the opinion of the Investigator, should undergo ventilatory (CPAP, mechanical ventilation, etc.) or circulatory support within 24 hours of study enrollment;
5. Have any serious acute concomitant illness that, in the opinion of the Investigator, would interfere with evaluation of safety or efficacy, or put the participant at risk of harm from study participation;
6. Are currently receiving an investigational agent, have participated in another study of an investigational agent within 30 days of enrollment, or were previously enrolled in the current study;
7. Are legally incompetent and unable to understand the study's purpose, significance, and consequences, and to make decisions accordingly;
8. Women who are pregnant or breast-feeding, or planning to conceive in the next 30 days;
9. Have known hypersensitivity to interferon alpha or any component of the study drug or placebo control.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 173 (Actual)
Dates: Start 2021-09-15 (Actual); Primary Completion 2022-04-15 (Actual); Study Completion 2022-07-28 (Actual)

PRIMARY OUTCOMES:
Treatment-emergent adverse events in healthy subjects | At the end of Phase 1 (Phase 1 is 11 days)
  Safety and tolerability of AP-003 as measured by subject incidence of treatment-emergent adverse events.
Change in perception of health status measured by EQ VAS in COVID-19 patients | At Day 5 of Phase 2 (Phase 2 is 28 days)
  Changes from baseline evaluation in COVID-19(+) participants' perception of health status at Day 5 as measured by EQ VAS in AP-003 treated patients compared to placebo.

SECONDARY OUTCOMES:
Serum levels of interferon alpha 2b | Up to Day 11 of Phase 1 (Phase 1 is 11 days)
  Pharmacokinetics of nebulized AP-003 in healthy adults assessed by serial serum quantification of interferon alpha 2b
Expression of interferon-induced genes in blood sputum samples | Up to Day 11 of Phase 1 (Phase 1 is 11 days)
  Evaluation of interferon-induced biomarkers after treatment with AP-003 in blood and sputum of healthy adults to assess biological effect of Interferon
Change in perception of health status measured by EQ VAS | Day 10 of Phase 2 (Phase 2 is 28 days)
  Changes in participants' perception of health status from baseline to Day 10 as measured by EQ VAS in AP-003 treated patients compared to placebo.
Change in perception of health status measured by EQ VAS | Day 28 of Phase 2 (Phase 2 is 28 days)
  Changes in participants' perception of health status from baseline to Day 28 as measured by EQ VAS in AP-003 treated patients compared to placebo.
Change in EuroQoL Quality of Life instrument (EQ-5D-5L) | Up to day 28 of Phase 2 (Phase 2 is 28 days)
  Changes in participants' perception of health status from baseline to Day 5, from baseline to Day 10, and from baseline to Day 28 as measured by EuroQoL Quality of Life instrument (EQ-5D-5L).
Change in Ordinal Scale for Clinical Improvement | Up to day 28 of Phase 2 (Phase 2 is 28 days)
  Changes in participants' overall health from baseline to Day 5, from baseline to Day 10, and from baseline to Day 28 as measured by Ordinal Scale for Clinical Improvement in AP-003 treated patients compared to placebo.
Improvement in clinical symptoms | Up to day 28 of Phase 2 (Phase 2 is 28 days)
  Changes in participant's improvement in clinical symptoms from baseline to Day 5, from baseline to Day 10, and from baseline to Day 28 as measured by a daily symptom diary in AP-003 treated patients compared to placebo.
Emergency department visits | Up to day 28 of Phase 2 (Phase 2 is 28 days)
  The proportion of participants attending an emergency department for COVID-19 by Day 28 in AP-003 treated patients compared to placebo.
Hospitalizations | Up to day 28 of Phase 2 (Phase 2 is 28 days)
  The proportion of participants hospitalized for COVID-19 by Day 28 in AP-003 treated patients compared to placebo.
Duration of hospitalization | Up to day 28 of Phase 2 (Phase 2 is 28 days)
  For hospitalized participants, duration of hospitalization in AP-003 treated patients compared to placebo.
Time from consent to clinical deterioration | Up to day 28 of Phase 2 (Phase 2 is 28 days)
  Time from consent to clinical deterioration defined as requiring or recommended for ventilatory support (continuous positive airway pressure [CPAP] or ventilator), shock requiring vasopressor support, and/or heart failure (defined as left ventricular ejection fraction [LVEF] < 30%) in AP-003 treated patients compared to placebo.
Change in SARS CoV-2 viral load | Up to day 28 of Phase 2 (Phase 2 is 28 days)
  SARS CoV-2 viral load by quantitative PCR from baseline to Day 5, from baseline to Day 10, and from baseline to Day 28 in AP-003 treated patients compared to placebo.
Change in inflammatory parameters | Up to day 28 of Phase 2 (Phase 2 is 28 days)
  Changes in D dimer, CRP, Ferritin, Troponin, creatine phosphokinase (CPK), LDH, IL-6 from baseline through Day 28 in AP-003 treated patients compared to placebo.
Organ failure rate | Up to day 28 of Phase 2 (Phase 2 is 28 days)
  Organ failure, any organ, from consent through Day 28 in AP-003 treated patients compared to placebo.
Death rate | Up to day 28 of Phase 2 (Phase 2 is 28 days)
  Death, any cause, from consent through Day 28 in AP-003 treated patients compared to placebo.

CONTACTS AND LOCATIONS:
Overall Officials: Arturo Borzutzky, M.D., Study Director — Pontificia Universidad Catolica de Chile; Diego García-Huidobro, M.D., Ph.D., Principal Investigator — Pontificia Universidad Catolica de Chile; Carolina Iturriaga, R.N., Principal Investigator — Pontificia Universidad Catolica de Chile; Jose A Castro-Rodríguez, M.D., Ph.D., Principal Investigator — Pontificia Universidad Catolica de Chile; Eleanor Fish, Ph.D., Principal Investigator — University Health Network, Toronto, Canada
Locations (1):
- Red de Salud UC Christus, Santiago, RM, Chile

IPD SHARING:
Plan to Share IPD: Yes
Available upon reasonable request.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Data will become available 1 year after study completion during 5 years upon reasonable request.
Access Criteria: Available upon reasonable request.

REFERENCES:
- [Derived] Garcia-Huidobro D, Iturriaga C, Perez-Mateluna G, Fajuri P, Severino N, Urzua M, Fraga JP, de la Cruz J, Poli C, Castro-Rodriguez JA, Fish E, Borzutzky A; IN(2)COVID Research Team. Safety, Tolerability, Bioavailability, and Biological Activity of Inhaled Interferon-alpha2b in Healthy Adults: The IN2COVID Phase I Randomized Trial. Clin Drug Investig. 2023 Jun;43(6):447-461. doi: 10.1007/s40261-023-01278-3. Epub 2023 Jun 22. PMID 37347370